CLINICAL TRIAL: NCT01588587
Title: Effect of DPP-IV Inhibitors on Occurence of Cancers and the Mechanism Using AGE and RAGE in Patients With Type 2 Diabetes
Brief Title: DPP-IV Inhibitors Underlying Mechanism of Cancer in Diabetic Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nagaoka Red Cross Hospital (Other)
Collaborators: Kurume University (Other)
Responsible Party: Principal Investigator, Kyuzi Kamoi, Medical Doctor, Nagaoka Red Cross Hospital
Other Study IDs: 7-Kamoi
Record Dates: First submitted 2012-04-26; First posted 2012-05-01 (Estimated); Last update posted 2012-10-19 (Estimated); Status verified 2012-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; alogliptin; Vildagliptin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- DPP-IV inhibitors
  Interventions: Drug: Sitagliptin; Drug: Alogliptin; Drug: Vildagliptin

INTERVENTIONS:
Drug: Sitagliptin — The dosage, frequency and duration for each sitagliptin are variant.
  Other Names: Other names are not known.
Drug: Alogliptin — The dosage, frequency and duration for each alogliptin are variant.
  Other Names: Other names are not known.
Drug: Vildagliptin — The dosage, frequency and duration for each vildagliptin are variant.
  Other Names: Other name is not known.

SUMMARY:
Recently, DPP-IV inhibitors are used as a novel way to augment the incretin system and one of the newest classes of medications in the treatment of type 2 diabetes mellitus (T2DM). Since the DPP-IV inhibitor was first used, about 5 years have passed in USA. However, there were no major side effects including occurrence of cancers. The main mechanism for DPP-IV inhibitors is due to suppress the function of DPP-IV activity. As it is known that the suppressed DPP-IV activity is a marker for early diagnosis of cancers, the reason of disassociation is not clear.

Activation of receptor for advanced glycation endproduct (AGE) is related to sideration of cancers. Meanwhile, the DPP-IV inhibitors may be related to inhibit the activation of receptor for AGE (RAGE). Therefore, DPP-IV inhibitors may work as a cancer protective agent in diabetes by blocking the AGE-RAGE axis.

However, it is not demonstrated why DPP-IV inhibitors have no side effect of occurrence of cancer via blocking the activation of AGE-RAGE.

The investigators examined effect of DPP-IV inhibitors on frequency of cancers and the underlying mechanism using AGE and RAGE before and 5 years after administration of DPP-IV inhibitors in Japanese patients with T2DM.

DETAILED DESCRIPTION:
The AGE and RAGE are measured using ELISA method in the laboratory of Department of Pathophysiology and Therapeutics of Diabetes Vascular Complications, Kurume University, School of Medicine, Japan before and for 5 years after administration of DPP-IV inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus patients with or without cancer

  * Patients who have no treatment with DPP-IV inhibitors.
  * Outpatients regularly visiting hospital
  * Patients 20 years old (gender is disregarded)

Exclusion Criteria:

* Patients with a serious complication in the heart, liver or kidney

  * Pregnant or possibly pregnant patients, or lactating patients
  * Patients participating in other clinical study.
  * Other than the above, patients judged inappropriate as the subjects of this study by the investigator

Ages: 20 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 500 patients
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2012-10; Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of cancers | Each one year within 5 years

SECONDARY OUTCOMES:
AGE concentration | Before and each one year within 5 years
  Serum AGE is measured using ELISA at the laboratory of Department pf Pathophysiology and Therapeutics of Diabetes Vascular Complications, Kurume University, which requre as 0.75 ml of serum in each patient.
Receptor for AGE concentration | Before and each one year within 5 years
  Serum receptor for AGE is measured using ELISA at the laboratory of Department pf Pathophysiology and Therapeutics of Diabetes Vascular Complications, Kurume University, which requre as 0.75 ml of serum in each patient

CONTACTS AND LOCATIONS:
Overall Officials: Kyuzi Kamoi, MD, Principal Investigator — Nagaoka Red Cross Hospital
Locations (2):
- Japan (2):
  - Kurume University, Kurume, Fukuoka
  - Nagaoka Red Cross Hospital, Nagaoka, Niigata

REFERENCES:
- [Result] 1.Gooβen K, Gräber S. Longer-term safety of DPP-4 inhibitors in patients with type 2 diabetes mellitus: systematic review and meta-analysis. Diabetes Obes Metab 2012 doi:[Epub ahead of print]. 2.Cornell S. Differentiating among incretin therapies: a multiple-target approach to type 2 diabetes. J Clin Pharm Ther 2012; 21:1365-2710. 3.Cordero OJ, Imbernon M, Chiara LD, Martinez-Zorzano VS, Ayude D, de la Cadena MP, Rodriguez-Berrocal FJ.Potential of soluble CD26 as a serum marker for colorectal cancer detection. World J Clin Oncol 2011;2: 245-61. 4.Taguchi A, Blood DC, del Toro G, Canet A, Lee DC, Qu W, Tanji N, Lu Y, Lalla E, Fu C, Hofmann MA, Kislinger T, Ingram M, Lu A, Tanaka H, Hori O, Ogawa S, Stern DM, Schmidt AM. Blockade of RAGE-amphoterin signalling suppresses tumour growth and metastases. Nature 2000;18;405:354-60.5.Kang R, Loux T, Tang D, Schapiro NE, Vernon P, Livesey KM, Krasinskas A, Lotze MT, Zeh HJ 3rd. The expression of the receptor for advanced glycation endproducts (RAGE) is permissive for early pancreatic neoplasia. Proc Natl Acad Sci U S A 2012 Apr 16. [Epub ahead of print].6.Ishibashi Y, Matsui T, Takeuchi M, Yamagishi S. Sitagliptin augments protective effects of GLP-1 against advanced glycation end product receptor axis in endothelial cells. Horm Metab Res 2011; 43:731-4.